CLINICAL TRIAL: NCT00385554
Title: Phase I Trial of the Safety, Toxicity, and Acceptability of the Microbicide UC-781 When Topically Applied by HIV-uninfected Women and Men in Botswana
Brief Title: Botswana Study of UC-781 Vaginal Microbicide
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study product is no longer being considered for further development.
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: CONRAD (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDC-NCHSTP 4885; BOTUSA MB05
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2012-08-16 (Estimated); Status verified 2012-08

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV prevention; Botswana; Preventing acquisition of HIV infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: UC-781 carbomer gel, 0.1% and 0.25%

SUMMARY:
This study will test the safety, side effects, and acceptability of two strengths of UC-781 gel when used by women and men in Botswana for two weeks.

DETAILED DESCRIPTION:
45 women and 45 men, all healthy and sexually active, 21-45 years old, without HIV infection, will be enrolled in Francistown and Gaborone, Botswana. Volunteers will be randomized to receive either 0.1% or 0.25% UC-781 carbomer gel or placebo gel (3 arms. Women will be instructed to apply gel intravaginally, morning and evening, and prior to sex (always with male condom use) for 14 consecutive days. Men will be instructed to apply gel topically for 14 consecutive nights, before bed, allow to dry overnight, and wash it off in the morning. Additionally instructed never to use gel during sex but always to use condoms. Volunteers will be seen weekly for evaluation of symptoms, laboratory toxicities, genital exam findings (with colposcopy for women, and plasma drug levels. Acceptability will be assessed in focus groups in the month after completing gel use.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years old
* citizen of Botswana
* willing to use condoms for 14 days
* PAP smear (normal, inflammation, ASCUS)
* regular menses or amenorrhea
* lives within 1 hour of a study clinic
* pass comprehension test
* provide written informed consent

Exclusion Criteria:

* genital mucosal disruption at screening
* genital surgery within past 8 weeks
* pregnant within past 8 weeks
* currently breastfeeding
* prior hysterectomy
* plans to move within 2 months
* ALT, AST, total bilirubin, or creatinine Grade 2 or above
* Prothrombin or partial thromboplastin time Grade 2 or above
* In other drug/vaccine safety trial
* Has more than one sexual partner in past month
* Unwilling/unsure they can have sex at least twice weekly for 2 weeks
* Any other condition that investigator believes will interfere with the evaluation of study objectives

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The safety and toxicity of 0.1% and 0.25% UC-781 carbomer gel compared to placebo gel in HIV uninfected, sexually active women and men

SECONDARY OUTCOMES:
Effects on vaginal microflora
Systemic absorption
Use acceptability in trial populations

CONTACTS AND LOCATIONS:
Overall Officials: Dawn K Smith, MD, MPH, Principal Investigator — BOTUSA/CDC; Christine K Mauck, MD, MPH, Study Director — CONRAD
Locations (3):
- United States (2):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - CONRAD, Arlington, Virginia
- BOTUSA HIV Prevention Research Unit, Gaborone and Francistown, Botswana